CLINICAL TRIAL: NCT01883154
Title: The Impact of Placental Factors on Fetal Intrauterine Growth and in Intrauterine Programming of the Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: loe135673ctil
Record Dates: First submitted 2013-06-11; First posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Normal Pregnancies

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — placental tissue ,fetal cord blood and maternal blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- IUGR pregnancies: Pregnancies complicated with IUGR. Fetal growth beneath the 10th percentile
- pregnancies with Gestational Diabetes: Normal glucose levels before 20 weeks, and positive Oral glucose tolerance test
- Pre Gestational Diabetes: A diagnosis of Diabetes before pregnancy or elevated glucose levels before 20 weeks.
- IVF pregnancies

SUMMARY:
Genetic and environmental factors are believed to play a major role in intrauterine growth and intrauterine programming. We intend to study genetic factors such as Telomere homeostasis, senescence, genomic instability and the presence of Genomic copy number variations in placental tissue from pregnancies complicated with Intrauterine growth restriction(IUGR), Gestational and pre gestational Diabetes, placentas from IVF pregnancies and from normal pregnancies. We also intend to assess these factors in cord blood and maternal blood.

DETAILED DESCRIPTION:
Based on the previous data from our group as well as other laboratories, we postulate that there is a correlation between impaired telomere homeostasis, senescence genomic instability and intra-uterine programming in placentas and in fetuses exposed to suboptimal intrauterine conditions such as hypoxia or hyperglycemia. Improved understanding of the mechanisms that produce the genomic changes in IUGR placentas and their influence on later risks of developing the metabolic syndrome should provide basis for future research that might lead into improved outcome of IUGR fetuses.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Intrauterine growth restriction
* A diagnosis of Gestational diabetes
* A diagnosis of pre gestational Diabetes
* IVF pregnancy

Exclusion Criteria:

* chorioamnionitis
* meconium stained amniotic fluid
* A request of the patient for Cord blood retrieval for preservation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Samples from pregnancies complicated with IUGR, Gestational and pre gestational Diabetes, placentas from IVF pregnancies and from normal pregnancies. We intend to assess these factors in placental tissue, in cord blood and maternal blood.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Copy Number Variations | 10 yeras

SECONDARY OUTCOMES:
Telomere length | 10 years
Number of copies of mitochondrial DNA | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center, Kfar Saba, Israel